CLINICAL TRIAL: NCT02793804
Title: Self-testing for HIV (HIVST) Amongst Urban, Peri-urban and Rural Communities in Zambia, Including a Cluster-randomised Trial of Community-based HIVST Distribution
Brief Title: HIV Self-Testing Africa Zambia
Acronym: STAR Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Zambart (Other); Society for Family Health, Zambia (Unknown); Liverpool School of Tropical Medicine (Other); University College, London (Other); Population Services International (Other); World Health Organization (Other); UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10660
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2017-08

CONDITIONS: HIV
Keywords: HIV self-testing; HIV; Zambia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): All HIV testing and counselling services will be conducted as currently.
- HIV Self-Testing (Experimental): Community-based distribution agents (CBDA), including Voluntary Male Medical Circumcision (VMMC) mobilisers, will deliver OraQuick® HIV Self-Tests (Orasure Technologies, Thailand). The kits will also be available at the health facility.
  Interventions: Device: Oraquick (made in Thailand)

INTERVENTIONS:
Device: Oraquick (made in Thailand)
  Arms: HIV Self-Testing

SUMMARY:
This study consists of a Cluster Randomised Trial (CRT) of community and facility-based HIVST distribution by the Society for Family Health (SFH) in multiple rural and peri-urban settings. The study will take place in 6 matched pairs of health facilities and their catchment areas have been selected for study inclusion in collaboration with the district medical office (DMO). One clinic catchment area from each pair will be randomly allocated to the HIVST arm (intervention) and the other to the standard of care (SOC) arm (Control).In the HIVST arm, community-based distribution agents (CBDA), including Voluntary Medical Male Circumcision (VMMC) mobilisers, will deliver HIVST kits. The kits will also be available at the health facility. In the SOC arm, all HIV testing and counseling (HTC) services will be conducted as currently.

DETAILED DESCRIPTION:
The study will use the OraQuick® HIV Self-Test (Orasure Technologies, Thailand). The kits contain the HIV Oral Fluid Test (HIVOFT) test kit, stand, buffer solution, locally-translated instructions for use (IFUs), materials on counselling and linkage to care, and primary and secondary packaging. The kits will be distributed for free by CBDAs. Leaflets will be provided in lieu of patient information sheets, but no other consent will be required for HIVST implementation.

Following baseline enumeration, clinic pairs will be randomly allocated to either the intervention or control arm at a public ceremony. An opaque bag containing 2 balls - one for HIVST and one for SOC - will be used to allocate the HIVST arm.

It will not be possible to blind participants, CBDAs, or their supervisors to the cluster intervention allocation, but all forms will be managed without reference to the intervention arm. Outcome data will not be analysed until completion of the trial, with the exception of data analysis by an independent statistician for presentation to the Trial Advisory Group.

CBDAs linked to intervention clinics will be provided with training in HIVST and Information, Education and Communication (IEC) materials including flipcharts, used kits to show clients how to interpret positive, negative and inconclusive results, a cotton bud and vial of water to demonstrate the mouth swabbing and development process, leaflets and a buffer stock of OraQuick® HIV Self-Test to be stored in a locked container in their own home.

Older adolescent and adult participants (age 15 - 17years or older) wishing to know their status will be provided with information on where to obtain further counselling and care together with the kit, and an envelope for return of the used kit, a self-completed questionnaire (SCQ), a self-referral slip for the nearest clinic in case of a positive result, and information on how to access VMMC for HIV-negative men.

Clients will be encouraged to return their used kits confidentially to the CBDA, either in person or by posting in the sealed envelope into an opaque locked "ballot box" container kept in/at the CBDA's/counsellor's house. Clients will also be encouraged to seek post-test advice from the CBDA, which can be "generic" or results-based.

Kits will be replaced by the clinic supervisors on presentation of used kits and following inspection of an HIV test logbook to confirm recording of names and addresses, but not results, of clients. Numbers of used kits, and re-read results, will be recorded by the CBDA/clinic supervisor. HIVST logbooks will be kept at the CBDA's home in a locked container. Couple's testing will be encouraged. In the case of couples wanting to self-test together, both partners will be asked to attend the IEC session. Clients will be allowed to take up to 2 kits home if the partner cannot attend. Testing of children (aged 15 years or less) will not be permitted as part of this trial, but can be arranged through special arrangement with SFH supervisors.

There are no sharps or hazardous materials that will be used in this study.

BASELINE SURVEY SAMPLING AND INCLUSION/EXCLUSION CRITERIA

Sample size calculations

Baseline enumeration will include approximately 2400 participants in the intervention communities (400 per community) and 2,400 participants in the control communities (n=~4,800). Within this sample, 20% of participants (~1,000) will be randomly selected for the extended baseline survey. The sample size justification for the extended questionnaire is detailed below.

The sample size was calculated to ensure 80% power to detect a 50% change in the proportion of individual tested for HIV over the last twelve months, with 95% confidence. Using 2013-2014 Demongraphic and Health Survey (DHS) data, baseline rates for individuals tested in the last 12 months are estimated to be between 28.6-57.1% (lower in men than women); for this sample calculation, we have assumed a baseline testing rate of 50%. For a two-sample comparison of matched proportions across 6 pairs of matched communities, we estimate that it will be necessary to recruit around 400 respondents per community, or 4,800 respondents in total.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Adolescents (16 and 17 years old)
* Able and willing to provide informed consent
* Residing within catchment area of a designated local health unit
* Residing in a randomly selected household

Exclusion Criteria:

* Unable and unwilling to provide informed consent
* Residing outside the catchment area.
* Anything that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5005 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison between randomisation arms in coverage of recent (within the last 12 months) HIV testing among older adolescents and adults (aged from 16 years) in the clinic catchment areas 12 months after the start of the intervention - by self-report | 12 months
  Recent testing will be measured by self-report and analyzed at the individual level. Respondents will be asked to answer the following question: "Have you tested for HIV within the past 12 months" as part of the baseline, midline, and endline surveys.

SECONDARY OUTCOMES:
Comparison between randomisation arms of antiretroviral therapy (ART) initiation rates for older adolescent and adult (aged from 16 years) cluster residents, during months 1 to 12 of the intervention - measured using clinic data | 12 months
  Linkage to HIV care will be measured using clinic data. Self-testers will receive self-referral forms, and will be asked to bring these to clinics where they receive confirmatory testing and care. Clinic staff will log all clients seeking confirmatory testing following HIV self-testing. Data on linkage will be aggregated to the clinic level for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Lusaka, Lusaka, Zambia

REFERENCES:
- [Derived] Neuman M, Hensen B, Mwinga A, Chintu N, Fielding KL, Handima N, Hatzold K, Johnson C, Mulubwa C, Nalubamba M, Otte Im Kampe E, Simwinga M, Smith G, Tsamwa D, Corbett EL, Ayles H. Does community-based distribution of HIV self-tests increase uptake of HIV testing? Results of pair-matched cluster randomised trial in Zambia. BMJ Glob Health. 2021 Jul;6(Suppl 4):e004543. doi: 10.1136/bmjgh-2020-004543. PMID 34275868
- [Derived] Neuman M, Indravudh P, Chilongosi R, d'Elbee M, Desmond N, Fielding K, Hensen B, Johnson C, Mkandawire P, Mwinga A, Nalubamba M, Ncube G, Nyirenda L, Nyrienda R, Kampe EOI, Taegtmeyer M, Terris-Prestholt F, Weiss HA, Hatzold K, Ayles H, Corbett EL. The effectiveness and cost-effectiveness of community-based lay distribution of HIV self-tests in increasing uptake of HIV testing among adults in rural Malawi and rural and peri-urban Zambia: protocol for STAR (self-testing for Africa) cluster randomized evaluations. BMC Public Health. 2018 Nov 6;18(1):1234. doi: 10.1186/s12889-018-6120-3. PMID 30400959